CLINICAL TRIAL: NCT03401866
Title: Multi-site Validation and Application of a Consensus Dynamic Susceptibility Contrast Magnetic Resonance Imaging (DSC-MRI) Protocol
Brief Title: Multi-site Validation and Application of a Consensus DSC-MRI Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-DSC-MRI-Quarles
Record Dates: First submitted 2017-12-11; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Glioblastoma Multiforme; Gliosarcoma
Keywords: brain tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DSC-MRI scan (Other): All subjects will receive a double dose injection protocol that will be split into multiple doses for sequential DSC-MRI scans.
  Interventions: Diagnostic Test: DSC-MRI

INTERVENTIONS:
Diagnostic Test: DSC-MRI — The multiple dose protocol with sequential DSC-MRI scans enables comparison of BTIP compliant and double-dose injections schemes."

SUMMARY:
This clinical trial is to validate and demonstrate the clinical usefulness of a protocol for Magnetic Resonance Imaging (MRI) in people with high grade glioma brain tumors.

DETAILED DESCRIPTION:
Although DSC-MRI itself is not novel, the consensus protocol tested herein is newly developed in response to a stated need by federal agencies (FDA, NCI) for standardization of imaging endpoints, including perfusion-weighted MRI, in multi-center clinical trials of GBM therapies. Through use of stereotactic methodologies that have been used to demonstrate that rCBV(relative cerebral blood flow) and FTB(fractional tumor burden) measures made by the consensus DSC-MRI protocol are concordant with tissue histology, this multi-site trial will be the first to validate a consensus DSC-MRI protocol on multiple platforms representing all major MRI scanner manufacturers. The trial also formally compares two contrast agent dosing schemes proposed in the consensus protocol, a single-dose BTIP-compliant scheme and a double-dose scheme. Such a comparison has never been tested in patients before, and addresses a longstanding controversy regarding contrast agent administration and dosing for DSC-MRI. Successful validation of the consensus DSC-MRI protocol will likely shift clinical practice paradigms. To date, the widespread adoption of DSC-MRI has been limited by inconsistent published methodologies, rCBV thresholds, and impact on clinical decision making. This trial seeks to improve confidence in DSCMRI methodology as it will foster its adoption for multicenter trials, facilitating the development and testing of novel therapeutic agents and treatment strategies for GBM, and shift clinical practice paradigms by providing strong evidence to support the inclusion of DSC-MRI in established response assessment criteria (i.e., modified RANO).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven intracranial glioblastoma or gliosarcoma at initial surgery
* Patient is currently being treated with standard first-line therapy for glioblastoma/gliosarcoma
* Karnofsky performance status ≥ 70
* Age ≥ 18 years
* Women must not be pregnant or breast-feeding as gadolinium enhanced MRI is contra-indicated
* Progressive contrast enhancement (> 25% increase in contrast enhancing volume compared to nadir, not corresponding to a region of peri-operative infarct seen on immediate post-op MRI) identified on routine surveillance MRI, with plan for surgical biopsy/resection. Measurable enhancement is defined as two perpendicular in-plane diameters of at least 10 mm and at least 10 mm in the 3rd orthogonal direction. This must be the patient's initial recurrence.
* Intratumoral hemorrhage (acute, subacute, or chronic) as seen on hemosiderin-sensitive (gradient-echo) MRI may preclude patient inclusion because of anticipated limited evaluation due to magnetic susceptibility artifact on the heavily T2*-weighted DSC-MRI images. If the region of enhancing tumor not affected by blooming artifact on the hemosiderin-sensitive images does not meet the 10 x 10 x 10 mm "measurable enhancement" threshold specified elsewhere, the patient is ineligible.
* Patients must be able to tolerate brain MRI scans with dynamic intravenous gadolinium-based contrast agent injections
* No known allergy-like reaction to gadolinium or moderate or severe allergic reactions to one or more allergens as defined by the American College of Radiology (ACR);
* Weight compatible with limits imposed by the MRI scanner table.

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Histologic measures of tumor fraction | 1 day
  Apply fractional tumor burden (FTB) rCBV thresholding methods to quantify recurrent tumor burden and compare this against histopathologic tumor burden from corresponding surgical specimens.

SECONDARY OUTCOMES:
Determine the repeatability of rCBV measured with the consensus DSC-MRI protocol. | 1 week
  "The repeatability of rCBV measured with the consensus DSC-MRI protocol will be quantified using the intra-class correlation coefficient (ICC).
Determine overall survival (OS) in recurrent GBM patients. | 3 years
  follow up for up to 3 years post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Chad Quarles, PhD, Principal Investigator — Barrow Neurological Institute
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Brown University, Providence, Rhode Island
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No